CLINICAL TRIAL: NCT01888237
Title: Randomized Open Labeled Clinical Trial: a Comparative Study of 10-day High Dose PPI-based Triple Therapy vs. 10-day Sequential Therapy for Helicobacter Pylori Eradication in Functional Dyspepsia Patients
Brief Title: High Dose PPI Triple Therapy Versus Sequential Therapy for Helicobacter Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Takeda Pharmaceuticals International, Inc. (Industry)
Responsible Party: Principal Investigator, Monthira Maneerattanaporn, Lecturer, Mahidol University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: si111/2013
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Dyspepsia; Helicobacter-associated Gastritis; Stomach Disorders
Keywords: Dyspepsia; Helicobacter pylori; Clarithromycin resistance; Other Specified Disorders of Function of Stomach
MeSH Terms: conditions — Dyspepsia; Stomach Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequential therapy (ST) (Active Comparator): 10 day Sequential therapy: lansoprazole 30 mg b.d. plus amoxicillin 1000 mg b.d. for 5 days then lansoprazole 30 mg b.d., metronidazole 400 mg b.d. and clarithromycin 500 mg b.d. for the remaining 5 days
  Interventions: Drug: sequence of drug use
- High dose PPI triple therapy(TT) (Experimental): 10 day high dose PPI triple therapy: lansoprazole 60 mg b.d. plus clarithromycin 500 mg b.d. and amoxycillin 1000 mg b.d. for 10 days
  Interventions: Drug: Double dose of PPI

INTERVENTIONS:
Drug: Double dose of PPI — Lansoprasole (30mg) 2 tab oral BID
  Arms: High dose PPI triple therapy(TT)
Drug: sequence of drug use — lansoprazole 30 mg b.d. for 10 days amoxicillin 1000 mg b.d. (day 1 to day 5) metronidazole 400 mg b.d. (day 6-day 10) and clarithromycin 500 mg b.d. (day 6-day 10)
  Arms: Sequential therapy (ST)

SUMMARY:
The purpose of this study is to compare the efficacy between 1-day high dose PPI-based triple therapy vs. 10-day sequential therapy for Helicobacter pylori eradication in functional dyspepsia patients.

DETAILED DESCRIPTION:
Background:

Helicobacter pylori (HP) play an important role in the pathogenesis of chronic gastritis, peptic ulcer diseases as well as gastric cancer. Helicobacter pylori eradication is a critical strategy to reduce aforementioned conditions. Proton-pump inhibitor (PPI)-based triple therapy (Standard dose PPIs+ Clarithromycin 1g/D + Amoxycillin 2g/D or Metronidazole 800 mg/D) is recommended as a frontline treatment in current guidelines for HP eradication, both from Thai and Second Asia-Pacific Consensus Guideline for H.pylori 2009. Unfortunately, it has been reported an unacceptably low eradication rate (<85%) of this regimen in a tertiary care hospital in Thailand. This occurrence is not surprised as the worldwide efficacy of this regimen had decreased to 50-75%. Of this, Clarithromycin resistance has been a major cause of the treatment failure.

Sequential therapy (ST) which consists of standard dose PPIs + amoxycillin 2 g/D for 5 days with 5 additional days of clarithromycin 1g/D + metronidazole 800 mg/D has been proposed to increase an efficacy in HP eradication. A recent meta-analysis of over three thousand population revealed a higher eradication rate over PPI-based triple therapy (TT). A consistent finding from Thailand was reported an impressive success rate of ST in HP eradication up to 95%. Therefore, more updated guidelines recommend using ST, not TT, as the first line regimen. However, ST is a complicated regimen for the patients to be followed. This might cause a low adherence rate in clinical practice as well as development of drug resistance in near future.

Interestingly, PPI is a pivotal in all regimens in HP eradication. There is evidence that the sustained higher intragastric pH is a major therapeutic determinant of HP eradication. Other factors including inflammatory cytokine polymorphisms, especially the IL-1B-511 T/T genotype and PPIs metabolizer, are the determinants of eradication by affecting gastric acid secretion and mucosal inflammation. Hence, higher dosage of PPIs is justified to eradicate HP. This has been shown in a recent meta-analysis that high dose PPI is better than standard dose PPI triple therapy in HP eradication of HP. Our study aims to compare the efficacy of ST to high dose PPI TT. Secondary outcomes include comparisons in the adherence and adverse events between both regimens, to determine the prevalence of clarithromycin resistance HP and determine improvement of dyspeptic symptoms after HP eradication

Primary Aim/Objective:

To evaluate eradication rates of Helicobacter pylori infection in functional dyspepsia patients amongst Thai population, compare between a 10-day sequential regimen (lansoprazole 30 mg b.d. plus amoxicillin 1000 mg b.d. for 5 days then lansoprazole 30 mg b.d., metronidazole 400 mg b.d. and clarithromycin 500 mg b.d. for the remaining 5 days) with a 10-day high dose PPI-based triple regimen (lansoprazole 60 mg b.d. plus clarithromycin 500 mg b.d. and amoxycillin 1000 mg b.d. for 10 days)

ELIGIBILITY:
Inclusion Criteria:

* Functional dyspepsia patients (Rome III) with rapid urease test positive
* Age ≥ 18 years old
* No history of HP eradication

Exclusion Criteria:

* Recent use of PPI, H2RA, NSAID, Antibiotics within 2 weeks
* Currently use of anticoagulants or ketoconazole
* C/I for gastric biopsy
* History of gastric surgery
* Comorbidity: ESRD, advanced cirrhosis, AIDS, stroke (bed ridden)
* Pregnancy or lactation
* Allergy to studied drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Eradication rate | 4 weeks after the end of intervention

SECONDARY OUTCOMES:
Adherence rate/adverse events | up to 2 weeks after intervention initiation
Prevalence of clarithromycin resistance HP | 4 weeks after the end of intervention
Symptomatic responses regarding dyspeptic symptoms after HP eradication | Baseline, week 4,8 and 24 after intervention completion

CONTACTS AND LOCATIONS:
Overall Officials: monthira maneerattanaporn, Principal Investigator — Division of gastroenterology, Department of Medicine, Siriraj hospital 2, Pran-nok, Bangkoknoi, Bangkok, Thailand, Mahidol University
Locations (1):
- Division of gastroenterology, Department of Medicine, Siriraj hospital, Bangkok Noi, Bangkok, Thailand

REFERENCES:
- [Derived] Auesomwang C, Maneerattanaporn M, Chey WD, Kiratisin P, Leelakusolwong S, Tanwandee T. Ten-day high-dose proton pump inhibitor triple therapy versus sequential therapy for Helicobacter pylori eradication. J Gastroenterol Hepatol. 2018 Nov;33(11):1822-1828. doi: 10.1111/jgh.14292. Epub 2018 Jun 27. PMID 29804294